CLINICAL TRIAL: NCT03177759
Title: Evaluating a Group Therapy Intervention to Alleviate Psychological Distress in Men With Prostate Cancer: An Assessment of a Group Therapy Program From Vancouver's Prostate Cancer Supportive Care (PCSC) Program
Brief Title: Living With Prostate Cancer (LPC)
Acronym: LPC
Status: Completed | Type: Observational
Sponsor: Vancouver Prostate Centre (Other)
Responsible Party: Sponsor
Other Study IDs: PCSC-6
Record Dates: First submitted 2017-03-07; First posted 2017-06-06 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective evaluation to determine the effectiveness of the Prostate Cancer Supportive Care (PCSC) Program's group therapy program, Living with Prostate Cancer (LPC). LPC is an intervention which utilizes a small group format (5-7 participants with 2 leaders and a paraprofessional counselling student) to understand and learn how to manage emotional responses, depressive symptoms, and life stressors associated with prostate cancer. Data for this evaluation will be derived from a focus group (at 3 months) and self-report questionnaires that participants will complete immediately prior to the intervention, immediately following the intervention and at 3, 6, and 12-months post-intervention.

DETAILED DESCRIPTION:
The Vancouver Prostate Centre's (VPCs) PCSC Program is designed to address the gap in supportive care for men with prostate cancer (PC), their partners and their families. The evaluation protocol described here is specific to the program called "Living with Prostate Cancer" (LPC) from the Psychooncology module of the PCSC Program. The specific rationale for this module is that many cancer patients will experience significant anxiety or depression at some point along their cancer journey. The module includes private, confidential clinic appointments for PC patients and their spouses/partners, either separately or together, with our registered clinical counsellor, to explore how to cope with difficult emotions such as fear, anxiety, sadness, helplessness, and other signs of emotional distress. The module is now being expanded to include small group discussions. LPC is a group therapy program in which men participate in a guided autobiographical life review through a process that focuses on developing a cohesive working group, learning strategic communication skills, and understanding and learning how to manage difficult emotions and transitional life stressors associated with PC. It also focuses on the processing and integrating of critical events that contribute to the men's present day identity and psychological function and involves the consolidation of the personal learning that occurs. It shifts the focus on transitioning into the future by developing specific individual, family and/or career goals that are reinforced by ongoing support from peers in the group. Finally, post-group referral plans are developed on an individual basis as needed.

The group therapy program includes men with a diagnosis of PC Stages 1 to 3. We will administer validated quantitative tools to assess depression and anxiety, general psychological functioning, and male role norms (masculinity) before, after, and at 3, 6, and 12-months following the program. The meeting 3 months after the program will include a focus group process.

ELIGIBILITY:
Inclusion Criteria:

Men are eligible to participate in this evaluation if they:

* are older than 18 years old
* are willing to attend the "Living with Prostate Cancer" group therapy sessions from the PCSC Program*
* are able to speak and read English such that they are able to understand the questionnaires
* have unimpaired cognitive function with an ability to understand the nature of the study
* are willing to complete questionnaires at 5 time points
* provide written informed consent

  * to be able to participate in LPC groups, men must have recently received a diagnosis of PC Stages 1 to 3, or have recently been recommended to undergo a form of treatment following a period of active surveillance.

Exclusion Criteria:

Men will be ineligible to participate in this evaluation if they:

* have difficulties reading or understanding English
* have psychotic symptoms, current severe alcohol or other drug dependence, unwillingness to refrain from substance use during the program, and/or significant cognitive impairment that would prevent them participating or providing full informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The LPC Workshops will only include men with a diagnosis of Prostate Cancer Stages 1 to 3.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in depressive and anxiety symptoms | Baseline (pre-workshop), 3-Weeks (Post-workshop), 3-, 6- and 12 Months
  Measured by the Beck Depression Inventory

SECONDARY OUTCOMES:
Changes in overall well-being | Baseline (pre-workshop), 3-Weeks (Post-workshop), 3-, 6- and 12 Months
  Measured by the Warwick-Edinburgh Mental Wellbeing Scale
Changes in perceptions of masculinity | Baseline (pre-workshop), 3-Weeks (Post-workshop), 3-, 6- and 12 Months
  Measured by the Personal Attributes Questionnaire
Changes in perceptions of masculinity | Baseline (pre-workshop), 3-Weeks (Post-workshop), 3-, 6- and 12 Months
  Measured by the Masculine Behaviour Scale
Group cohesion and dynamics | 3-Weeks (Post-workshop), 3-, 6- and 12 Months
  Measured by the Group Questionnaire
Patient-incurred costs for attending the session | 3-Weeks (Post-Workshop)
  Measured by an annotated cost questionnaire for completion by patients

CONTACTS AND LOCATIONS:
Overall Officials: David Kuhl, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Prostate Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No